CLINICAL TRIAL: NCT02158858
Title: A Phase 1/2 Study of CPI-0610, a Small Molecule Inhibitor of BET Proteins: Phase 1 (Dose Escalation of CPI-0610 in Patients With Hematological Malignancies) and Phase 2 (Dose Expansion of CPI-0610 With and Without Ruxolitinib in Patients With Myeloproliferative Neoplasms)
Brief Title: A Phase 1/2 Study of CPI-0610 With and Without Ruxolitinib in Patients With Hematologic and Myeloproliferative Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Constellation Pharmaceuticals (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0610-02; 2018-000579-34 (EudraCT Number); CDAK539A12201 (Other: Novartis)
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Myelofibrosis; Leukemia, Myelocytic, Acute; Myelodysplastic/Myeloproliferative Neoplasm; Myelodysplastic Syndrome (MDS); Preleukemia; Primary Myelofibrosis; Myeloproliferative Disorders; Bone Marrow Disease; Hematological Disease; Precancerous Conditions; Neoplasms; Leukemia; Neoplasms by Histologic Type; Essential Thrombocytosis
Keywords: Phase 1; Phase 2; Oncology; BET Inhibitor; Ruxolitinib; Pelabresib (CPI-0610)
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myeloid, Acute; Myelodysplastic-Myeloproliferative Diseases; Myelodysplastic Syndromes; Preleukemia; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; Precancerous Conditions; Neoplasms; Leukemia; Neoplasms by Histologic Type; Thrombocythemia, Essential | interventions — CPI-0610; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 (Experimental): Patients are enrolled in sequential cohorts (acute leukemia, including acute myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), and acute undifferentiated or biphenotypic leukemia; chronic myelogenous leukemia (CML) in blast crisis; myelodysplastic syndrome (MDS); myelodysplastic/myeloproliferative neoplasms (MDS/MPN); or myelofibrosis (MF)) and receive escalating doses of pelabresib (CPI-0610).
  Interventions: Drug: Pelabresib
- Phase 2 (Arm 1): Prior JAKi Monotherapy Arm (MF patients treated with pelabresib alone) (Experimental): * Cohort 1A: Open to patients with MF who are Transfusion Dependent (TD) and who have previously been treated with a JAKi and are intolerant, resistant, refractory or lost response to the JAKi, or are ineligible to be treated with a JAKi (pelabresib (CPI-0610) alone)
  * Cohort 1B: Open to patients with MF who are not TD and who have previously been treated with a JAKi and are intolerant, resistant, refractory or lost response to the JAKi, or are ineligible to be treated with a JAKi. (pelabresib (CPI-0610) alone)
  Interventions: Drug: Pelabresib
- Phase 2 (Arm 2): Prior JAKi Combination Arm (Experimental): * Cohort 2A: Open to patients with MF who are Transfusion Dependent (TD) and are currently taking ruxolitinib but have disease that is not being adequately controlled by ruxolitinib (pelabresib (CPI-0610) + Ruxolitinib)
  * Cohort 2B: Open to patients with MF who are not TD and are currently taking ruxolitinib but have disease that is not being adequately controlled by ruxolitinib. (pelabresib (CPI-0610) + Ruxolitinib)
  Interventions: Drug: Pelabresib; Drug: Ruxolitinib
- Phase 2 (Arm 3): JAKi Naïve Combination Arm (Experimental): Open to patients with MF who have not previously received a JAKi (pelabresib (CPI-0610) + Ruxolitinib)
  Interventions: Drug: Pelabresib; Drug: Ruxolitinib
- Phase 2 (Arm 4): Essential Thrombocythemia (ET) Monotherapy Arm (Experimental): Open to high-risk patients with ET who are resistant or intolerant to hydroxyurea (HU) (pelabresib (CPI-0610) alone)
  Interventions: Drug: Pelabresib

INTERVENTIONS:
Drug: Pelabresib — CPI-0610 is administered orally once daily for 14 consecutive days, followed by a 7-day break (1 cycle = 21 days)
  Other Names: CPI-0610; DAK539
Drug: Ruxolitinib — Ruxolitinib is given orally, twice daily (BID), on a continuous basis for 21 consecutive days of each 21-day cycle.
  Arms: Phase 2 (Arm 2): Prior JAKi Combination Arm; Phase 2 (Arm 3): JAKi Naïve Combination Arm

SUMMARY:
Phase 1 Part: Open-label, sequential dose escalation study of pelabresib (CPI-0610) in patients with previously treated Acute Leukemia, Myelodysplastic/Myeloproliferative Neoplasms, and Phase 2 Part: Open-label study of pelabresib (CPI-0610) with and without Ruxolitinib in patients with Myeloproliferative Neoplasms (Myelofibrosis and Essential Thrombocythemia).

Pelabresib (CPI-0610) is a small molecule inhibitor of bromodomain and extra-terminal (BET) proteins.

ELIGIBILITY:
Phase I (Dose Escalation) - Inclusion and Exclusion Criteria:

1. Inclusion Criteria (Phase I):

   * Age: Adults ≥18 years.
   * Diagnosis: Histologically or cytologically confirmed diagnosis of one of the following hematologic malignancies:

     * Acute myelogenous leukemia (AML)
     * Acute lymphocytic leukemia (ALL)
     * Acute undifferentiated or biphenotypic leukemia
     * Chronic myeloid leukemia (CML) in blast crisis
     * Myelodysplastic syndrome (MDS)
     * Myelodysplastic/myeloproliferative neoplasms (MDS/MPN)
     * Myelofibrosis (MF)
   * Performance Status: ECOG ≤2.
   * Organ Function:

     * Serum total bilirubin ≤1.5 × ULN
     * AST/ALT ≤2.5 × ULN (up to 5 × ULN if due to leukemic infiltration)
     * Serum creatinine ≤2.0 × ULN or CrCl ≥30 mL/min
   * Hematology (MF only):

     * Platelet count ≥50 × 10⁹/L and ANC ≥1 × 10⁹/L (MF not on ruxolitinib)
     * Platelet count ≥75 × 10⁹/L and ANC ≥1 × 10⁹/L (MF on ruxolitinib)
   * Other:

     * DIPSS-plus risk category of intermediate-2 or high (MF only)
     * Serum glucose ≤160 mg/dL (or HbA1C ≤7%)
     * Fully recovered from major surgery and acute toxic effects of prior therapy
     * Negative pregnancy test for women of childbearing potential
     * Agreement to use appropriate contraception
     * Written informed consent
2. Exclusion Criteria (Phase I):

   * Untreated newly diagnosed acute leukemia (unless AML with myelodysplasia-related changes and 20-30% blasts)
   * Relapsed/refractory acute leukemia where further induction chemotherapy is beneficial
   * Acute leukemia relapse <6 months after allogeneic SCT
   * CML in blast crisis treated with only one TKI
   * Very low/low risk MDS without prior treatment
   * CNS involvement by leukemia (unless resolved)
   * Active HIV, Hepatitis B or C infection
   * GI impairment affecting absorption (unresolved nausea, vomiting, diarrhea >CTCAE grade 1)
   * Significant cardiac disease (recent MI/angina, high cTn, QTcF >470 ms, LVEF <50%, uncontrolled arrhythmia, etc.)
   * Severe/uncontrolled comorbidities
   * Recent systemic anti-cancer therapy (other than hydroxyurea/radiotherapy) <2 weeks prior
   * Ongoing or recent JAK inhibitor use (<2 weeks prior, MF only)
   * Recent therapeutic antibody (<4 weeks) or investigational agent (<2 weeks or <5 half-lives)
   * Use of strong CYP450 inhibitors/inducers or drugs with Torsades de Pointes risk
   * Immunosuppressive treatment that cannot be discontinued
   * Pregnant/lactating women
   * Inadequate contraception
   * Inability/unwillingness to comply with protocol

Phase II (Expansion) - Inclusion & Exclusion Criteria:

1. Inclusion Criteria (Phase II):

   1. MF Arms (Prior JAKi, Add-on JAKi, JAKi Naïve)

      * Age: Adults ≥18 years
      * Diagnosis: Confirmed primary MF or MF evolved from ET or PV
      * Risk: DIPSS intermediate-2 or higher
      * Platelets:

        * ≥75 × 10⁹/L (Arms 1 & 2)
        * ≥100 × 10⁹/L (Arm 3, JAKi naïve)
      * ANC: ≥1 × 10⁹/L
      * Spleen Volume: ≥450 cm³ by MRI/CT (non-TD cohorts) OR
      * Transfusion Dependence: Average ≥2 RBC transfusions/month (total ≥6 in prior 12 weeks) for TD cohorts
      * Peripheral Blood Blasts: <10%
      * Symptoms: At least 2 symptoms measurable (score ≥1 for Arms 1 & 2; score ≥3 or total ≥10 for Arm 3) using MFSAF v4.0
      * Treatment History:

        * Arm 1 (Prior JAKi): Previously treated with JAKi and intolerant, resistant, refractory, or lost response, or ineligible for JAKi
        * Arm 2 (Add-on JAKi): On ruxolitinib ≥6 months, stable dose ≥8 weeks, not adequately controlled
        * Arm 3 (JAKi Naïve): No prior JAKi, eligible for ruxolitinib
      * Performance Status: ECOG ≤2
      * Organ Function: Serum direct bilirubin <2 × ULN, AST/ALT ≤2.5 × ULN (up to 5 × ULN if due to liver involvement), CrCl ≥45 mL/min
      * Other: Fully recovered from major surgery/acute toxic effects, effective contraception, written informed consent
   2. ET Arm (High-Risk ET)

      * Age: Adults ≥18 years
      * Diagnosis: Confirmed ET (WHO 2016 criteria)
      * High-Risk: At least one of:

        * Age >60 years
        * Platelets >1500 × 10⁹/L
        * Prior thrombosis, erythromelalgia, or migraine (disease-related)
        * Prior hemorrhage related to ET
        * Diabetes/hypertension requiring therapy >6 months
      * Symptoms: ≥2 symptoms with average score ≥3 or total score ≥15 (MPN-SAF)
      * Platelets: >600 × 10⁹/L
      * Resistant/Intolerant to HU: As defined by ELN
      * Performance Status: ECOG ≤2
      * Life Expectancy: >24 weeks
      * ANC: ≥1 × 10⁹/L
      * Organ Function: Serum direct bilirubin <2 × ULN, AST/ALT ≤2.5 × ULN, CrCl ≥45 mL/min
      * Other: Fully recovered from major surgery/acute toxic effects, effective contraception, written informed consent
2. Exclusion Criteria (Phase II)

   * Prior splenectomy (MF non-TD cohorts)
   * Splenic irradiation within 3 months
   * Active or chronic HIV, Hepatitis B/C infection
   * Active clinically significant infection (until recovery ≥2 weeks)
   * Anemia deemed clinically significant (iron/B12/folate deficiency, hemolytic anemia)
   * Major bleeding event (≥2 g/dL Hgb drop or ≥2 units transfused in last 6 months)
   * Liver cirrhosis Child-Pugh B or C
   * GI impairment affecting absorption (unresolved nausea, vomiting, diarrhea >CTCAE grade 1)
   * Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption (Arm 3)
   * Hypersensitivity to ruxolitinib formulation (Arm 3)
   * History of PML (Arm 3)
   * Significant cardiac disease (recent MI/angina, QTcF >500 ms [>450 ms in France/Germany], uncontrolled arrhythmia, etc.)
   * Ongoing uncontrolled hypertension
   * Severe/uncontrolled comorbidities
   * Systemic anticancer treatment (other than ruxolitinib for Arm 2, HU/ANA up to 24h prior) <2 weeks or <5 half-lives prior
   * Prior treatment with any BET inhibitor
   * Hematopoietic growth factor or androgenic steroids <4 weeks prior
   * Systemic corticosteroids ≥10 mg prednisone equivalent within 4 weeks (exceptions for short courses)
   * Concurrent/second malignancy (except certain adequately treated cancers)
   * Pregnant/lactating women, or planning pregnancy within protocol-defined window
   * Inability/unwillingness to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Phase 1: Frequency of Dose-limiting toxicities (DLTs) | DLTs assessed during Cycle 1 (cycle = 21 days)
  The maximum tolerated dose (MTD) of CPI-0610 and characterize its DLTs in patients with acute leukemia, myelodysplastic syndrome (MDS), myelodysplastic/myeloproliferative neoplasms (MDS/MPN), and myelofibrosis (MF), when given once daily by mouth for 14 consecutive days followed by a 7-day break.
Phase 2 (Cohorts 1B, 2B, and Arm 3): Splenic Response Rate by Imaging | 24 weeks (Cycle 9, Day 1)
  Splenic response rate is defined as the proportion of patients who achieve a ≥ 35% reduction from baseline spleen size by imaging (MRI or CT) after 24 weeks of treatment.
Phase 2 (Cohorts 1A and 2A): Conversion rate from Red Blood Cell (RBC) transfusion dependence (TD) to transfusion independence (TI) | 12 consecutive weeks (rolling window, assessed after 24 weeks)
  Conversion rate is defined as the proportion of patients who convert from TD to TI, where TD is defined as receiving an average of ≥ 2 units of RBC transfusions per month (total of ≥ 6 RBC transfusions during the 12 weeks) prior to enrollment and TI is defined as absence of RBC transfusions over any consecutive 12 week period
Phase 2 (Arm 4): Complete Hematological Response (CHR) Rate | Over 2 consecutive cycles (rolling window) (1 cycle = 21 days)
  Complete CHR rate is defined as the proportion of patients who meet the criteria for CHR, as assessed by modified European LeukemiaNet (ELN) criteria: platelet count ≤400 × 10⁹/L, WBC ≤10 × 10⁹/L, laboratory results confirmed after 1 cycle, and normal spleen size by palpation or imaging.

SECONDARY OUTCOMES:
Phase 1: Incidence rate of adverse events (AEs), serious adverse events (SAEs) | Through Phase I completion, an average of 4 years
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 4.03.
Phase 2 (All Arms): Incidence rate of adverse events (AEs), serious adverse events (SAEs) | Through Phase II completion, an average of 6 years
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 4.03.
Phase 2 (All Arms): Change from Baseline in Patient Global Impression of Change (PGIC) at 12 and 24 weeks | Baseline, 12 weeks (Cycle 5, Day 1), 24 weeks (Cycle 9, Day 1)
  The Patient Global Impression of Change (PGIC) is a single-question, patient-reported assessment that asks individuals to rate their overall change in myeloproliferative neoplasm (MPN) symptoms since starting study treatment. The patient select one of seven options, ranging from "Very much improved" to ""Very much worse". No Change from Baseline indicates stable symptoms (no improvement or worsening), negative change from Baseline indicates a reduction in symptom severity (improvement) and positive change from Baseline indicates an increase in symptom severity (worsening).
Phase 2 (Arms 1, 2 and 3): Change from Baseline in Myelofibrosis Symptom Assessment Form (MFSAF v4.0) at 12 and 24 weeks | Baseline, 12 weeks (Cycle 5, Day 1), 24 weeks (Cycle 9, Day 1)
  The MFSAF (Myelofibrosis Symptom Assessment Form) should be completed by patients every day for 7 days before Day 1 of each treatment cycle, including the 7 days before starting Cycle 1. It uses a 24-hour recall format, asking patients to rate the worst severity of seven symptoms (fatigue, night sweats, pruritus, abdominal discomfort, pain under the ribs on the left side, early satiety, and bone pain) during the past 24 hours. Each symptom is rated on a scale from 0 (Absent) to 10 (Worst Imaginable). The Total Symptom Score (TSS) is the sum of 7 symptoms (range: 0 - 70). No Change from Baseline indicates stable symptoms (no improvement or worsening), negative change from Baseline indicates a reduction in symptom severity (improvement) and positive change from Baseline indicates an increase in symptom severity (worsening).
Phase 2 (Arms 1, 2 and 3): Percentage of patients who achieve a ≥ 50% reduction in Total Symptom Score (TSS) at 12 and 24 weeks | 12 weeks (Cycle 5, Day 1), 24 weeks (Cycle 9, Day 1)
  The "percentage" of study participants whose TSS-measured by the Myelofibrosis Symptom Assessment Form (MFSAF v4.0)-decreases by at least half compared to their baseline score, when assessed at 12 weeks and again at 24 weeks.
Phase 2 (Arms 1, 2 and 3): Overall splenic response rate at 12 and 24 weeks | 12 and 24 weeks
  The overall splenic response rate is the proportion of patients who achieve a ≥ 35% reduction from baseline spleen size by imaging (MRI or CT).
Phase 2 (Arms 1, 2 and 3): Splenic response at 12 and 24 weeks | 12 and 24 weeks
  The reduction in spleen size from baseline by imaging (MRI or CT) after 12 weeks (Cycle 5, Day 1) and after 24 weeks of treatment (Cycle 9, Day 1) will also be evaluated.
Phase 2 (Arms 1, 2 and 3): Duration of Transfusion Independence (TI) | From first onset of TI to earliest onset of loss of TI, assessed up to approximately 6 years
  Time from first onset of TI to earliest onset of loss of TI.
Phase 2 (Arms 1, 2 and 3): Early anemic response rate | Through Phase II completion, an average of 6 years
  Proportion of patients who achieve a hemoglobin increase of ≥1 g/dL from baseline, without RBC transfusions.
Phase 2 (Arms 1, 2 and 3): Anemic response rate in TI patients | Through Phase II completion, an average of 6 years
  Proportion of TI patients with ≥1.5 g/dL hemoglobin increase from baseline, without RBC transfusions.
Phase 2 (Arms 1, 2 and 3): Duration of splenic response | From first onset of splenic response until loss of response, assessed up to approximately 6 years
  Time from first meeting splenic response criteria until loss of response (spleen volume <35% reduction from baseline and increased by ≥25% from nadir).
Phase 2 (Arms 2 and 4): Maximum observed plasma concentration (Cmax) of pelabresib and ruxolitinib | Cycle 1 Day 14 (30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 8 hours post-dose). 1 cycle = 21 days.
  Pharmacokinetic (PK) parameters will be calculated based on Pelabresib and Ruxolitinib plasma concentrations and actual sampling time points.
  Cmax will be listed and summarized using descriptive statistics.
Phase 2 (Arms 2 and 4): Time to reach maximum concentration (tmax) of pelabresib and ruxolitinib | Cycle 1 Day 14 (30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 8 hours post-dose). 1 cycle = 21 days.
  Pharmacokinetic (PK) parameters will be calculated based on Pelabresib and Ruxolitinib plasma concentrations and actual sampling time points.
  Tmax will be listed and summarized using descriptive statistics.
Phase 2 (Arms 2 and 4): Predose (trough) concentration at the end of a dosing interval (Ctrough) of pelabresib and ruxolitinib | Cycle 1 Day 1, Cycle 1 Day 14, Cycle 3 Day 1: predose. 1 cycle = 21 days.
  Pharmacokinetic (PK) parameters will be calculated based on Pelabresib and Ruxolitinib plasma concentrations and actual sampling time points.
  Ctrough will be listed and summarized using descriptive statistics.
Phase 2 (Arms 2 and 4): Area under the concentration-time curve from time zero to the last observed concentration (AUClast) of pelabresib and ruxolitinib | Cycle 1 Day 14 (30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 8 hours post-dose). 1 cycle = 21 days.
  Pharmacokinetic (PK) parameters will be calculated based on Pelabresib and Ruxolitinib plasma concentrations and actual sampling time points.
  AUClast will be listed and summarized using descriptive statistics.
Phase 2 (Arms 2 and 4): Area under the concentration-time curve from time zero to 8 hours post-dose at steady state (AUC0-8,ss) of pelabresib and ruxolitinib | Cycle 1 Day 14, Cycle 3 Day 1. 1 cycle = 21 days.
  Pharmacokinetic (PK) parameters will be calculated based on Pelabresib and Ruxolitinib plasma concentrations and actual sampling time points.
  AUC0-8,ss will be listed and summarized using descriptive statistics.
Phase 2 (Arms 2 and 4): Maximum concentration at steady state (Cmax,ss) of pelabresib and ruxolitinib | Cycle 1 Day 14, Cycle 3 Day 1. 1 cycle = 21 days.
  Pharmacokinetic (PK) parameters will be calculated based on Pelabresib and Ruxolitinib plasma concentrations and actual sampling time points.
  Cmax,ss will be listed and summarized using descriptive statistics.
Phase 2 (Arms 2 and 4): Time to reach maximum concentration at steady state (tmax,ss) of pelabresib and ruxolitinib | Cycle 1 Day 14, Cycle 3 Day 1. 1 cycle = 21 days.
  Pharmacokinetic (PK) parameters will be calculated based on Pelabresib and Ruxolitinib plasma concentrations and actual sampling time points.
  Tmax,ss will be listed and summarized using descriptive statistics.
Phase 2 (Arm 4): Percentage of patients who achieve a ≥50% reduction from baseline in the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) total score | Baseline, 12 weeks (Cycle 5, Day 1), 24 weeks (Cycle 9, Day 1)
  The Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) is a patient-reported questionnaire designed to measure symptom burden in patients with myeloproliferative neoplasms (MPNs). Patients rate the severity of several symptoms (such as fatigue, night sweats, itching, abdominal discomfort, bone pain, early satiety, and others) over the past 24 hours. Each symptom is scored on a scale from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be). The total score is the sum of all individual symptom scores, providing an overall measure of symptom burden. A 50% reduction in the MPN-SAF total score at 12 or 24 weeks means the patient's overall symptom burden has improved by half compared to their baseline (pre-treatment) score.
Phase 2 (Arm 4): Partial Hematological Response Rate | Over 2 consecutive cycles (rolling window) (1 cycle = 21 days)
  Proportion of patients with platelets 400-600 × 10⁹/L, WBC ≤10 × 10⁹/L, confirmed after 1 cycle.
Phase 2 (Arm 4): Overall Hematological Response Rate | Through Phase II completion, an average of 6 years
  Proportion of patients with complete or partial hematological response.
Phase 2 (Arm 4): Duration of Hematological Response | Through Phase II completion, an average of 6 years
  Time from first onset of response to earliest onset of loss of response, including hematologic response and symptom improvement
Phase 2 (Arm 4): Rate of hemorrhagic and thromboembolic (TE) events | Through Phase II completion, an average of 6 years
  Proportion of patients with hemorrhagic or TE events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (48):
- United States (12):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern University - Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Washington University School of Medicne Neuromuscular Division Department of Neurology Research, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Weill Medical College and New York Presbyterian Hospital, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - UZ Leuven - Campus Gasthuisberg, Leuven, Viaams Braban
  - AZ Sint-Jan Burgge-Oostende AV- Campus Sint-Jan, Bruges, West-Vlaanderen
  - ZNA Stuyvenberg Antwerpen, Antwerp
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (5):
  - Institut de cancérologie du Gard - Hematologie clinique, Nîmes, Gard
  - CHRU de Lille - Hopital Claude Huriez, Toulouse, Haute-Garonne
  - CHRU de Lille - Hopital Claude Huriez - Maladies du Sang, Lille, Hauts-de-France
  - CHU - Hopital Saint Louis - Centre D'Investigations Clinique, Paris
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Germany (2):
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
- Italy (8):
  - Institue of Hematology "L. and A. Seràgnoli", Bologna, Emilia-Romagna
  - Servizio Sanitario Regionale Emilia-Romagna - Azienda Unita Sanitaria Locale (AUSL) di Rimini - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - AOU S.Martino, IRCCS, IST-Istituto Nazionale Ricerca Sul Can, Genoa, Liguria
  - Ospedale Maggiore Policlinico, Fondazione IRCCS Ca' Granda, Milan, Lombardy
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia, Lombardy
  - Ospedale di Circolo, PO Varese, AO Ospedale di Circolo e Fon, Varese, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - AOU Maggiore della Carità, Novara
- Netherlands (3):
  - Maastricht University Medical Center, Maastricht, Limburg
  - VUmcResearch B.V., Amsterdam, North Holland
  - Erasmus Universitair Medisch Centrum Rotterdam, Rotterdam, South Holland
- Poland (2):
  - Instytut Hematologii i Transfuzjologii w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
- United Kingdom (8):
  - Oxford University Hospitals, Headington, Oxford
  - Belfast City Hospital, Belfast
  - University of Cambridge, Cambridge
  - University Hospital of Wales, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospital's NHS foundation Trust, London
  - Guys and St Thomas' Hospital - Haematology, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Stein EM, Fathi AT, Harb WA, Colak G, Fusco A, Mangan JK. Results from phase 1 of the MANIFEST clinical trial to evaluate the safety and tolerability of pelabresib in patients with myeloid malignancies. Leuk Lymphoma. 2024 Apr;65(4):503-510. doi: 10.1080/10428194.2023.2300710. Epub 2024 Jan 23. PMID 38259250
- [Derived] Gupta V, Mascarenhas J, Kremyanskaya M, Rampal RK, Talpaz M, Kiladjian JJ, Vannucchi AM, Verstovsek S, Colak G, Dey D, Harrison C. Matching-adjusted indirect comparison of the pelabresib-ruxolitinib combination vs JAKi monotherapy in myelofibrosis. Blood Adv. 2023 Sep 26;7(18):5421-5432. doi: 10.1182/bloodadvances.2023010628. PMID 37530627
- [Derived] Mascarenhas J, Kremyanskaya M, Patriarca A, Palandri F, Devos T, Passamonti F, Rampal RK, Mead AJ, Hobbs G, Scandura JM, Talpaz M, Granacher N, Somervaille TCP, Hoffman R, Wondergem MJ, Salama ME, Colak G, Cui J, Kiladjian JJ, Vannucchi AM, Verstovsek S, Curto-Garcia N, Harrison C, Gupta V. MANIFEST: Pelabresib in Combination With Ruxolitinib for Janus Kinase Inhibitor Treatment-Naive Myelofibrosis. J Clin Oncol. 2023 Nov 10;41(32):4993-5004. doi: 10.1200/JCO.22.01972. Epub 2023 Mar 7. PMID 36881782